CLINICAL TRIAL: NCT04701333
Title: Cabergoline for Lactation Inhibition After Second-Trimester Abortion or Loss
Acronym: LISTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 58470
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Lactation Suppressed
Keywords: abortion; intrauterine fetal demise; second-trimester; lactation; engorgement
MeSH Terms: conditions — Stillbirth; Breast Feeding; Hyperemia | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cabergoline (Experimental): After the completion of the surgical procedure or medical induction for the second-trimester abortion or fetal loss, the participant will be administered cabergoline 1mg orally with juice or water by the clinician or study investigator.
  Interventions: Drug: Cabergoline 1 MG
- Placebo (Placebo Comparator): After the completion of the surgical procedure or medical induction for the second-trimester abortion or fetal loss, the participant will be administered a placebo pill orally with juice or water by the clinician or study investigator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabergoline 1 MG — Dopamine agonist
  Other Names: Dostinex
  Arms: Cabergoline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This research study investigates the use of a drug, cabergoline, given immediately after second-trimester abortion or perinatal loss to decrease breast engorgement. Cabergoline is a medication approved for the symptomatic treatment of pituitary adenomas that result in a hyperprolactinemic state (a brain tumor that results in milk leakage). The benefit of stopping milk leakage has also been studied and used in populations who shouldn't breastfeed. The investigators aim to clarify if cabergoline is effective in preventing breast engorgement and milk leakage after second-trimester abortions or perinatal loss (stillbirth). Breast engorgement causes physical pain and emotional distress as lactation is uniquely associated with parenthood and those undergoing second-trimester abortions are doing so because they choose not to parent or a previously desired pregnancy is now complicated by anomalies. As there are no current recommendations for management of this painful engorgement beyond icepacks and support bras, the investigators aim to validate the use of this pharmacologic option in this setting.

DETAILED DESCRIPTION:
Breast pain following second-trimester abortion is common. Breast engorgement and milk leakage following second-trimester perinatal loss and abortion can cause both physical pain and emotional distress. Dopamine agonists have previously been shown to be effective in lactation inhibition for third-trimester fetal/neonatal loss or contraindications to breastfeeding. In a head-to-head trial, cabergoline was more effective with a better safety profile than bromocriptine and has thus emerged as preferred treatment for term lactation inhibition internationally. Despite the frequency of breast symptoms after second-trimester abortions, there are no current guidelines for this population.

The investigators are conducting a double-blinded, placebo-controlled, superiority trial of participants undergoing abortion or experiencing intrauterine fetal demise between 18 and 28-weeks gestation at Stanford Health Care. Participants will be randomized to either cabergoline 1mg or placebo the day of procedure. Participants will complete the Bristol Breast Inventory, a survey to assess symptoms and side-effects at baseline and day 2, 3, 4, 7, and 14 after the procedure.

The primary outcome is breast symptoms on Day 4 as reported on the Bristol Breast Inventory. Secondary outcomes include satisfaction, acceptability, and side-effects. Investigators hypothesize that cabergoline is superior to placebo for preventing breast engorgement after second-trimester abortion or loss. A sub-study of 6 participants will return for serum prolactin levels at baseline, days 4, 7, 14 after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people, ages 18 years or older
* Intrauterine pregnancy between 18/0-28/0 weeks of gestation age (by ultrasound dating performed prior to or same day of enrollment visit)
* Consented for an induced, elective abortion or undergoing induction for demise
* English or Spanish speaking
* Able to consent for a research study, literate in English or Spanish
* Willing to comply with study procedures and follow-up
* Access to smart phone throughout study

Exclusion Criteria:

* Prior mastectomy (breast reduction or chest masculinization surgery acceptable)
* Currently breastfeeding
* Currently receiving dopamine agonist therapy for other indication (prolactinoma, Cushings syndrome, acromegaly, restless leg syndrome)
* Contraindication to cabergoline (as per package insert)

  * Uncontrolled hypertension - defined as baseline BP > 150/100, or chronic hypertension requiring more than one baseline medication, or pregnancy-induced hypertension spectrum disorders (gestational hypertension, preeclampsia, eclampsia)
  * History of cardiac valvular disorders or valvular repair
  * History of pulmonary, pericardial, or retroperitoneal fibrotic disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be requested for meta-analysis inclusion.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Henkel A, Reeves MF, Shaw KA. The experience of breast symptoms after second-trimester abortion or pregnancy loss. Am J Obstet Gynecol. 2024 Mar;230(3):e3-e5. doi: 10.1016/j.ajog.2023.10.025. Epub 2023 Oct 18. No abstract available. PMID 37863161
- [Derived] Henkel A, Johnson SA, Reeves MF, Cahill EP, Blumenthal PD, Shaw KA. Cabergoline for Lactation Inhibition After Second-Trimester Abortion or Pregnancy Loss: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jun 1;141(6):1115-1123. doi: 10.1097/AOG.0000000000005190. Epub 2023 May 3. PMID 37486652

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabergoline | Placebo
Started | 36 | 37
Completed | 33 | 29
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 3 | 7
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabergoline | Placebo | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (5.4) | 31.6 (5.7) | 31.1 (5.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 35 | 37 | 72
  Non-binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 14 | 15 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 15 | 26
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 7 | 5 | 12
Gestational age at time of procedure [Mean (Standard Deviation); unit: days] | 148.9 (13.4) | 147.7 (12.8) | 148.3 (13.0)
Nulliparous [Number; unit: participants] | 16 | 25 | 41
Indication [Count of Participants; unit: Participants]
  Undesired pregnancy | 14 | 8 | 22
  Fetal anomaly | 20 | 27 | 47
  Maternal comorbidity | 0 | 1 | 1
  Fetal demise | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Breast Pain
Description: Participants will assess their breast symptoms using the validated Bristol Breast Inventory survey to assess 4 domains of breast symptoms: tenderness, engorgement, leaking milk, pain relief. Participants who indicated symptoms in any of these areas met the criteria for this outcome.
Time Frame: Day 4 after procedure
Population: Participants who returned survey data for this outcome are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 36 | 33
Participants | 10 | 32

2. Secondary Outcome: Number of Participants Experiencing Side-effects
Description: Participants selected from previously documented side-effects from the dopaminergic class or free-text. Participants may have reported more than one side-effect.
Time Frame: 2 weeks
Population: Participants who returned survey data for this outcome are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 36 | 36
Participants
  Nausea/ vomiting | 5 | 2
  Headache | 12 | 9
  Dizziness/ lightheadness | 7 | 7
  Constipation | 14 | 18
  Acid reflux | 3 | 2
  Fatigue | 12 | 11
  Lower extremity edema | 4 | 4
  Hot flashes | 2 | 9
  Palpitations | 1 | 1
  Anxiety | 4 | 3
  Insomnia | 8 | 11
  Visual disturbance | 1 | 2

3. Secondary Outcome: Number of Participants Reporting Significant Bother From Breast Pain
Description: Assessed using a Facial Pain Score (scale range 0-6, significant bother >=4)
Time Frame: Day 4 after procedure
Population: Participants who returned survey data for this outcome are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 36 | 33
Participants | 1 | 11

4. Secondary Outcome: Serum Prolactin Level
Description: A subset of participants returned blood tests to measure effectiveness of drug
Time Frame: Day 4 after procedure
Population: Participants who returned for serum blood draws
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 3 | 3
ng/mL | 6.5 (2.2) | 18.0 (5.9)

5. Secondary Outcome: Number of Participants Reporting Significant Bother From Side-effects
Description: Assessed using a Facial Pain Score (scale range 0-6, significant bother >=4)
Time Frame: Day 4 after procedure
Population: Participants who returned survey data for this outcome are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 36 | 33
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: From day of enrollment until 14 days after procedure
Arm/Group | Cabergoline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04701333/Prot_SAP_001.pdf